CLINICAL TRIAL: NCT03283033
Title: Salad Bars and Students' Fruit and Vegetable Consumption: A Group-randomized Trial With Objective Assessments
Brief Title: School Lunch Salad Bars and Fruit and Vegetable Consumption
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 closed schools in March 2020. Data collection for all elementary schools was completed pre-pandemic. For middle and high schools, the marketing phase was halted. Results will solely reflect the salad bar intervention.
Sponsor: Arizona State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Marc Adams, PhD, MPH, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL139120 (NIH)
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Children, Only; Behavior, Eating; School; Obesity; Food Selection; Food Habits; Diet Modification; Adolescent Behavior
Keywords: Children; Plate Waste; Fruit and vegetable intake; School lunch; social marketing
MeSH Terms: conditions — Feeding Behavior; Obesity; Food Preferences; Adolescent Behavior | interventions — Marketing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 3 (Experimental): Introduction of a new salad bar and marketing conditions during second semester of school year
  Interventions: Behavioral: New salad bar; Behavioral: Marketing
- Experimental 2 (Experimental): Introduction of marketing conditions during second semester of school year
  Interventions: Behavioral: Marketing
- Experimental 1 (Experimental): Introduction of a new salad bar during second semester of school year
  Interventions: Behavioral: New salad bar
- Control (No Intervention): No introduction of a new salad bar and no introduction of marketing conditions

INTERVENTIONS:
Behavioral: New salad bar — New salad bar placed in school
  Arms: Experimental 1; Experimental 3
Behavioral: Marketing — Marketing conditions (printed material, displays, verbal announcements, prompts and taste tests)
  Arms: Experimental 2; Experimental 3

SUMMARY:
The investigators propose an efficacy study (i.e., do salad bars work under controlled conditions in naturalistic settings) to test whether introducing salad bars in elementary, middle, and high schools that have never had salad bars affects students' FV consumption and waste during lunch. A cluster randomized controlled trial will test new salad bars against controls for 6 wks, with/without an additional 4-wk marketing phase .

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in any grade between grades one and twelve
* Student ID number matches that on a list of randomly selected student ID numbers from the population of student enrolled in school
* Students who elect to receive a hot entree at lunch
* Students who assent to participate

Exclusion Criteria:

* Students in detention
* Students in special education
* Students in Kindergarten
* Students not in school for any reason (e.g. illness, vacation)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7491 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in grams of fruit and vegetables consumed | Baseline (prior to randomization allocation of installation of salad bars), Time 2 (6 weeks after randomization), and Time 3 (10 weeks after randomization)
  The amount (grams) of fresh and canned fruits and vegetables consumed at lunch

SECONDARY OUTCOMES:
Change in grams of fruit and vegetables selected | Baseline (prior to randomization allocation of installation of salad bars), Time 2 (6 weeks after randomization), and Time 3 (10 weeks after randomization)
  The amount (grams) of fresh and canned fruits and vegetables selected at lunch
Change in percent of fruit and vegetables wasted | Baseline (prior to randomization allocation of installation of salad bars), Time 2 (6 weeks after randomization), and Time 3 (10 weeks after randomization)
  The percent of fresh and canned fruits and vegetables wasted at lunch

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams MA, Ohri-Vachaspati P, Richards TJ, Todd M, Bruening M. Design and rationale for evaluating salad bars and students' fruit and vegetable consumption: A cluster randomized factorial trial with objective assessments. Contemp Clin Trials. 2019 Feb;77:37-45. doi: 10.1016/j.cct.2018.12.007. Epub 2018 Dec 18. PMID 30572161
- [Result] Bruening M, Adams MA, Ohri-Vachaspati P, Hurley J. Prevalence and Implementation Practices of School Salad Bars Across Grade Levels. Am J Health Promot. 2018 Jul;32(6):1375-1382. doi: 10.1177/0890117116689159. Epub 2017 Feb 19. PMID 29214812
- [Derived] Adams MA, Todd M, McEntee ML, Yu TY, Ohri-Vachaspati P, Richards TJ, Bruening M. A cluster randomized factorial trial of school-lunch salad bars and marketing on elementary students' objectively measured fruit and vegetable consumption. Int J Behav Nutr Phys Act. 2025 May 26;22(1):58. doi: 10.1186/s12966-025-01758-z. PMID 40420203